CLINICAL TRIAL: NCT02110433
Title: Heart Failure Educational and Follow up Platform
Acronym: HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHRD0414; 2013A0089936 (Other: IDRCB)
Record Dates: First submitted 2014-03-07; First posted 2014-04-10 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; BNP; telemedicine; telemonitoring; weight; education; self management; cost effectiveness
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo group (Other): Patients will be managed per consensus guidelines Clinicians could see the patients as many times as necessary in order to optimize their therapy and could make BNP measurement (but not using Home BNP monitoring)
  Interventions: Device: Placebo group
- Cordiva System (R) (Experimental): Patient will see their cardiologist every three months and benefit from telemonitoring of their weight and general well being through a specific communicant device.
  Interventions: Device: Cordiva System (R)
- BNP and Cordiva (R) monitoring system (Active Comparator): In this group, patients and doctors have access to the platform detailed above (Cordiva (R) monitoring system) and had also access to BNP home monitoring (BNP heartcheck).
  Interventions: Device: Cordiva System (R); Device: BNP heartcheck

INTERVENTIONS:
Device: Placebo group — patient will be managed as recommended by ESC guidelines and follow up will be in accordance to ESC recommendations
  Arms: Placebo group
Device: Cordiva System (R) — Patients have to answer to 8 specific binary questions based on the main precipitating factors for decompensation and measure their body weight every day. If not they will be contact after two missing measures. Patient will be contact by phone call every month in order to reinforce the initial patient therapeutic education and patient-'s compliance. Patient have access to specific printed documents and to a specific web based platform where he can find some PowerPoint presentation on CHF aetiology, signs and therapy and where he can try to answer to monthly quiz in whom questions are based on key messages about CHF according to guidelines and consensus paper on patient therapeutic education.
  Arms: BNP and Cordiva (R) monitoring system; Cordiva System (R)
Device: BNP heartcheck — Patients had to measure the BNP plasma level using Alere home based BNP device heartcheck in a weekly basis in order to follow this parameter up. In case of clinical signs of CHF or a significant weight increase identified by the tele monitoring or the patient, the nurse will ask to the patient to do an extra measurement of home BNP testing in order to exclude a CHF decompensation (BNP < 100 pg/ml or remaining stable (< 30% increase).
  Arms: BNP and Cordiva (R) monitoring system

SUMMARY:
Heart failure is a serious and common disease. HF is marked by a high rate of preventable hospitalizations through proper care. As such, it is a key target for telemedicine programs. However, currently published data are inconclusive. Investigators propose a multicenter randomized study of innovative telemedicine involving the usual patient monitoring daily weight monitoring, clinical signs and in one of three groups in our study of BNP testing in the patient's home all associated with a regular education reinforcement. The objective is to identify early cardiac decompensation to allow to treat ambulatory and thus prevent the occurrence of more serious events such as death or rehospitalization.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a disease that has several specificities. It is both common and severe. This is a disease associated with high mortality and especially a high rate of hospitalization. These are partly due to the severity " per se "of the disease but also to the non optimal management of CHF and non-formal education of patients and their caregivers. Indeed, the majority of hospitalized patients shows some clinical signs of decompensation up to 5 days before hospitalization and could avoid to go to the emergency room and hospitalization by an adequate ambulatory reaction and care. It is on this premise that underlies the concept of the application of telemedicine in CHF. Telemedicine is the monitoring of biological or clinical data in the patient's home with the transfer of information remotely either to a specific structure often managed by nurses or to the GP or cardiologist.

In most studies of telemedicine, effectiveness of the concept is based on the notion of monitoring of some markers with low sensitivity or specificity. This monitoring generates a lot of information which, because of the better education of the patient and from its systematic examination or through technology (internet, phone, SMS) or through remote monitoring of the nurse often leads to detection of sources of unnecessary hospitalization and offset the advantage gained in the early detection of decompensation. In addition, the low sensitivity and specificity of clinical signs generate many warnings that cause difficult remote management by the patient and the doctor. BNP is a blood biomarker recognized as having a high negative predictive value for the diagnosis of CHF and the rate change was correlated with a change in the prognosis. Its dosage is conventionally performed in peripheral blood using POCT devices or not. More recently, it is possible to perform the dosage by the patient itself at home, including a satisfactory feasibility.

This is why, in the HELP study , Investigators wanted to study the impact of the addition of BNP measurement at patient's home to a innovative device for telemedicine monitoring combining patient perception of clinical signs of HF decompensation, daily weight monitoring and strengthening patient education but also specific training of doctors by E learning in order to promote implementation of the ESC recommendations.

Study hypotheses

The primary objective of the HELP study is to determine the impact of a tele monitoring strategy based on either a telemonitoring of the weight associated with an educational reinforcement (clinical monitoring arm) or on the same track associated with a BNP assay at home performed by the patient every week and in case of symptoms suggestive of decompensation (bioclinical monitoring arm) on a primary endpoint including death from all causes, unscheduled re-hospitalization or CHF admission to the emergency department compared to a control group (usual monitoring arm).

Be secondarily analyzed the impact in terms of re-hospitalizations, deaths emergency admissions, the number of false positives (unconfirmed suspected cardiac decompensation), false negatives (undetected cardiac decompensation), the effect of monitoring quality of life and economic impact of these medical strategies.

Study design, inclusion, and exclusion criteria HELP (n° ansm 2013-A00899-36 ) is a multicentric, prospective, open label, randomized, ambulatory study. The authors are solely responsible for the design and conduct of this study, all study analyses, the drafting and editing of the paper, and its final contents. HELP study benefit form a specific grant of the Ile de France regional health agency, France. The aim was to initially include 330 patients suffering from ambulatory CHF according to inclusion and exclusion criteria Study procedures Patients should be followed by the study investigators. After signing the informed consent (approval by a French legal ethical committee on 8 th October 2013 N° 2013-A00899-36-3101), patients will be randomized into three arms according to their type of CHF (systolic CHF and CHF with preserved systolic function defined by the coexistence of signs of CHF and an ejection fraction> 45%). Patients will therefore be included into a standard of care arm (placebo group), one arm followed by clinical and telemonitoring arm ( Cordiva System (R) arm) followed by bio-clinical monitoring (BNP and Cordiva (R) monitoring system arm) . Patients will be seen per protocol at inclusion and 3, 6, 9 and 12 months after inclusion.

* Placebo arm group: Patients will be managed per consensus guidelines Clinicians could see the patients as many times as necessary in order to optimize their therapy and could make BNP measurement (but not using Home BNP monitoring)
* Cordiva System (R) arm : Patient will see their cardiologist every three months and benefit from telemonitoring of their weight and general well being through a specific communicant device. Patients have to answer to 8 specific binary questions based on the main precipitating factors for decompensation and measure their body weight every day. If not they will be contact after two missing measures. Patient will be contact by phone call every month in order to reinforce the initial patient therapeutic education and patient-'s compliance. Patient have access to specific printed documents and to a specific web based platform where he can find some PowerPoint presentation on CHF aetiology, signs and therapy and where he can try to answer to monthly quiz in whom questions are based on key messages about CHF according to guidelines and consensus paper on patient therapeutic education. The cardiologist has access to a specific platform. In this platform they could find the E CRF of their patients and the patient 's quiz result in order to help him to analyse patient comprehension of HF and patient reactivity in case of decompensation. The cardiologist could also find some PowerPoint presentation on CHF and AHF management according to ESC guidelines. He could also read the monthly report of the telemonitoring nurse and the daily results of weight and general being measurement of his patients.
* BNP and Cordiva (R) monitoring system arm : In this group, patients and doctors have access to the platform detailed above and had also access to BNP home monitoring. Patients had to measure the BNP plasma level using Alere home based BNP device heartcheck in a weekly basis in order to follow this parameter up. In case of clinical signs of CHF or a significant weight increase identified by the tele monitoring or the patient, the nurse will ask to the patient to do an extra measurement of home BNP testing in order to exclude a CHF decompensation (BNP < 100 pg/ml or remaining stable (< 30% increase).

End Points

Primary end point is a composite end point including Unplanned hospitalizations for CHF with hospital stay > 1 day / all-cause death / non-programmed emergency department admission related to CHF.

Secondary endpoint are based on an analysis of the impact of the strategy used in the two interventional arms compared to the placebo group for:

* each parameter of the composite end point analyzed separately
* emergency admission.
* Number of all cause death.
* Number of HF hospitalizations
* Patient management
* Adherence to the strategy
* Quality of life.
* False positive induced by the system (visits to the GP or cardiologist proposed by the telemonitoring system without final evidence of HF decompensation and without increase of diuretics )
* Medical cost and efficience of the technique
* Cost of the different strategies
* Cost efficacy of the different strategies

Hospitalization for heart failure was defined per protocol by an in-hospital stay of more than one night in addition with intravenous use of diuretics.

Statistical analysis Events in the three groups were analyzed using parametric student t test. Percentages were compared using Chi2 tests. Kaplan Meier time to event function for readmission or death from any cause were calculated. For each end point, investigators also estimated the hazard ratio and 95% confidence interval using a Cox proportional-hazards To calculate sample size, analyzing recent clinical trial data, investigators expected at least 40% of SOC subjects will have at least one cardiovascular event within 1 year. Assuming a 40% reduction in the occurrence of the primary end point in the telemonitoring groups , investigators estimated that a sample size of at least 110 subjects in each group would provide 80% power (α = .05) for detection of a reduction in primary end point. An initial goal enrollment of 330 subjects was proposed. According to the event rate in the control group study size could be secondarily extended to 600 patients.

Sub group analysis Actual prespecified sub group analysis were defined according to some patients characteristics or locations : Investigators also tested for interactions between each pair of subgroups and the main treatment effect.

Age (cut off 65 y old ) and above and below median value. PSEF versus REF (defined by EF > 45%) aetiology of CHF as defined by the investigator High symptomatic patients vs low symptomatic patients according to NYHA class Heart failure units management (defined by the investigator as working in such a structure) vs all others High neurohormonal activation patients vs low neurohormonal activation defined as initial BNP higher or lower than 300 pg/ml and in an second analysis by median initial BNP value.

patient adherence to the " phone call system " (<75% vs. ≥75%) BNP Compliant vs non compliant patients defined by an compliance to daily measurement plus BNP measurement in BNP group higher than 80%.

Highly implicated vs low implication patients defined according to the monthly connection to the patient site and median value during the study.

Good HF education level vs low HF education patients defined by tertile value of quiz performance (global, knowledge and situation questions as isolated value).

ELIGIBILITY:
Inclusion Criteria:

* Heart failure diagnosed on a first hospitalization for acute exacerbation during the last twelve months, without high age limit
* Men or women
* More than 18 years old
* Minimal knowledge of the French language (patient or his relatives)
* The patient need to fill an informed written consent
* Patient resides or is treated in Ile de France
* Patient is insured under the social security system

Exclusion Criteria:

* Myocardial infarction or revascularization or Heart Valve Surgery < 3 months
* Inability to execute the feasibility test
* Major cognitive disorders do not allow access to the platform
* Patient does not have the necessary autonomy to use the equipment
* Sensitive subject, under Article L32 of the Code of Public Health
* Patient enrolled in another clinical trial
* Renal failure with creatininemia clearance (cockcroft) <15 ml/min
* 24h/day oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Primary end point is a composite end point including unplanned hospitalizations for CHF with hospital stay > 1 day / all-cause death / non-programmed emergency department admission related to CHF | Follow up 12 months after inclusion
  Unplanned hospitalizations for CHF with hospital stay > 1 day / all-cause death / non-programmed emergency department admission related to CHF

SECONDARY OUTCOMES:
Number of emergency admission. | 12 months
  Count of emergency admission.
Number of all cause death. | 12 months
  Count of all cause death.
Number of HF hospitalizations | 12 months
  Count of HF hospitalizations
Adherence to the strategy | 12 months
  defined with at least 75% of the measurements done by the patient
Evaluation of life quality . | 12 months
  Use of eq-5d-3l at 3, 6, 9 and 12 month. In this questionnaire, 0 is the worst imaginable health state and 100 is the best imaginable health state
Number of false positive induced by the system (visits to the GP or cardiologist proposed by the telemonitoring system without final evidence of HF decompensation and without increase of diuretics ) | 12 months
  Visits to the GP or cardiologist proposed by the telemonitoring system without final evidence of HF decompensation and without increase of diuretics
Number of false positive induced by the system | 12 months
  Visits to the GP or cardiologist proposed by the system without final evidence of need
Cost of the different strategies | 12 months
  cost of hospitalization reported in the national health cost system / cost of transportation / cost of medical therapy (oral) / cost of medical visits / cost of the heartcheck monitoring system as mentioned by Alere(R)
Cost efficacy of the different strategies | 12 months
  cost of hospitalization reported in the national health cost system / cost of transportation / cost of medical therapy (oral) / cost of medical visits / cost of the heartcheck monitoring system as mentioned by Alere(R)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick JOURDAIN, Principal Investigator — René Dubos Hospital (Pontoise-France)
Locations (15):
- France (15):
  - Victor Dupouy Hospital, Argenteuil
  - Sud francilien Hospital, Corbeil-Essonnes
  - Henri-Mondor Hospital, Créteil
  - Simone Veil Hospital, Eaubonne
  - Bernard Clinic, Ermont
  - Gonesse Hospital, Gonesse
  - Versailles Hospital, Le Chesnay
  - Orsay Hospital, Longjumeau
  - Meaux Hospital, Meaux
  - Sainte Marie Clinic, Osny
  - Georges Pompidou University Hospital, Paris
  - Mutualiste Montsouris Institute, Paris
  - Turin Clinic, Paris
  - Poissy-Saint-Germain-en-Laye Hospital, Saint-Germain-en-Laye
  - Centre Hospitalier René DUBOS, Pontoise, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558